CLINICAL TRIAL: NCT02825459
Title: Does Abstinence From E-cigarettes Produce Withdrawal Symptoms?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Hughes, Faculty, Department of Psychiatry, University of Vermont
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01CA192940-01 (NIH); R01CA192940-01 (NIH)
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Substance Withdrawal Syndrome
Keywords: abstinence; abuse liability; electronic cigarette; e-cigarette; electronic nicotine delivery device; harm reduction; nicotine; nicotine dependence; smoking; smoking cessation; tobacco; vape; vaping; withdrawal
MeSH Terms: conditions — Substance Withdrawal Syndrome; Vaping; Harm Reduction; Tobacco Use Disorder; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abstinence from e-cigarettes (Experimental): Participants abstain from e-cigarettes and other nicotine/tobacco products for 6 days
  Interventions: Behavioral: Abstinence from e-cigarettes
- E-cigarette use (No Intervention): Participants use e-cigarettes and continue to abstain from tobacco/nicotine products as they normally would.

INTERVENTIONS:
Behavioral: Abstinence from e-cigarettes — Abrupt cessation for 6 days
  Arms: Abstinence from e-cigarettes

SUMMARY:
The purpose of this study is to see whether adults who use e-cigarettes every day experience symptoms of nicotine withdrawal when they stop using e-cigarettes for 6 days.

DETAILED DESCRIPTION:
Study Design: The investigators will recruit 120 individuals who are long-term daily and exclusive users of nicotine-containing e-cigarettes. Participants will be asked to use their own e-cigarette as usual during the first week of the study and to then stop their use of e-cigarettes for 6 days. The total study duration will be 14 days. Participants will be instructed to continue abstinence from other tobacco and nicotine products during the entire study. The investigators will use an escalating payment system with bonuses based on breath and urine samples to encourage compliance.

Every day during the study, participants will report e-cigarette and tobacco cigarette use and monitor symptoms of nicotine withdrawal via a phone call to an Interactive Voice Response system. Participants will attend 3 study visits each week to provide urine and breath samples to verify compliance, and to complete brief surveys.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to read and understand verbal English fluently
* US citizen or resident alien
* Primarily uses e-cigarette product types of refillable tanks or modified devices
* Uses nicotine-containing e-liquid
* Has baseline urinary cotinine concentration of > 100 ng/ml
* Has used e-cigarettes daily for the last 2 months
* Has a home or cell phone
* Agrees to abstain from tobacco, marijuana and other illegal drugs during study

Exclusion Criteria:

* Smoked > 5 tobacco cigarettes in the last month
* Used non-cigarette nicotine, tobacco or quit smoking products on >5 days in the past month
* Use of cannabis (either marijuana or synthetic cannabis) > 5 times in the past month or positive test for cannabis use at screening
* Current (last 6 months) Generalized Anxiety Disorder, Major Depressive Disorder, Attention Deficit Hyperactivity Disorder or moderate/severe Substance Abuse Disorder
* Multiple legal, social health, work or school problems in the past month due to alcohol or drug use
* Pregnant or breastfeeding
* Previously a participant in the current study
* Use of prescribed or non-prescribed psychoactive medication > 5 times in the past month
* Expired carbon monoxide level > 8ppm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-07; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Total score on the Minnesota Nicotine Withdrawal Scale (MNWS) | 6 days
  The investigators will compare the mean score across participants for the entire 6-day abstinence vs. use conditions.

SECONDARY OUTCOMES:
Individual items on the Minnesota Nicotine Withdrawal Scale (MNWS) | 6 days
  The investigators will use the mean score for each of the 16 symptoms across participants during abstinence and use conditions.
Questionnaire of E-cigarette Urges (brief) | 6 days
  This is a revision of the brief version Questionnaire of Smoking Urges that asks about urges for e-cigarettes rather than tobacco cigarettes.
Questionnaire of Smoking Urges- brief version | 6 days
  This 2-item scale asks about intensity and frequency of urges.
Heart rate | 6 days
  Measured for 30 sec after sitting for 15 minutes
E-cigarette Purchase Task | 6 days
  This is a modification of the Cigarette Purchase Task that asks how much users would expend to obtain their usual amount of e-liquids to use.

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Battelle Memorial Institute, Baltimore, Maryland
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes JR, Peters EN, Callas PW, Peasley-Miklus C, Oga E, Etter JF, Morley N. Withdrawal Symptoms From E-Cigarette Abstinence Among Adult Never-Smokers: A Pilot Experimental Study. Nicotine Tob Res. 2020 Apr 21;22(5):740-746. doi: 10.1093/ntr/ntz169. PMID 31504882
- [Derived] Hughes JR, Peters EN, Callas PW, Peasley-Miklus C, Oga E, Etter JF, Morley N. Withdrawal Symptoms From E-Cigarette Abstinence Among Former Smokers: A Pre-Post Clinical Trial. Nicotine Tob Res. 2020 Apr 21;22(5):734-739. doi: 10.1093/ntr/ntz129. PMID 31352486